CLINICAL TRIAL: NCT05795608
Title: Effectivity of Incentive Spirometry on Postoperative Pulmonary Complication After Major Abdominal Surgery In Indonesia Three Major Tertiary Hospitals: A Randomized Controlled Trial
Brief Title: Effectivity of Incentive Spirometry on Postoperative Pulmonary Complication After Major Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Cipto Mangunkusumo General Hospital (Other)
Responsible Party: Principal Investigator, Ridho Ardhi Syaiful, Medical Doctor, Digestive Surgery, Dr Cipto Mangunkusumo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RSyaiful
Record Dates: First submitted 2023-03-21; First posted 2023-04-03 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Incentive Spirometry; Postoperative Pulmonary Complication; Major Abdominal Surgery
Keywords: Incentive spirometry; major abdominal surgery; pulmonary complication

STUDY DESIGN:
Intervention Model Description: Subjects in the intervention group were trained to perform 15 minutes of respiratory exercise with incentive spirometry four times a day for two days before surgery by trained medical personnel. First, subjects were instructed to make a good seal over the incentive spirometry mouthpiece with their lips. Afterward, they were asked to inhale deeply and slowly, and they were also directed to hold their breath at the end of inspiration.
Who Masked: Investigator
Oversight: FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): The intervention group received respiratory exercise with incentive spirometry before surgery
  Interventions: Device: respiratory exercise with incentive spirometry
- control group (No Intervention): The control group were given standard preoperative care.

INTERVENTIONS:
Device: respiratory exercise with incentive spirometry — Subjects in the intervention group were trained to perform 15 minutes of respiratory exercise with incentive spirometry four times a day for two days before surgery by trained medical personnel. First, subjects were instructed to make a good seal over the incentive spirometry mouthpiece with their lips. Afterward, they were asked to inhale deeply and slowly, and they were also directed to hold their breath at the end of inspiration
  Arms: intervention group

SUMMARY:
This study is the first clinical trial study in Indonesia to assess the benefits of using incentive spirometry in the incidence of pulmonary complications after major abdominal surgery.

This study was a randomized clinical trial in three tertiary-level referral hospitals in Indonesia (Cipto Mangunkusumo Hospital, Fatmawati Hospital, and Persahabatan Hospital). The investigators randomly assigned adult patients who underwent major abdominal elective surgery in July-August 2015 to two groups.

All study subjects were simple randomly allocated to the intervention and control groups according to the randomization table.

The hypothesis of the study team was that preoperative incentive spirometry can improve the incidence of postoperative pulmonary complications in major abdominal surgery

DETAILED DESCRIPTION:
This study was a randomized clinical trial in three tertiary-level referral hospitals in Indonesia (Cipto Mangunkusumo Hospital, Fatmawati Hospital, and Persahabatan Hospital). The researchers randomly assigned adult patients who underwent major abdominal elective surgery in July-August 2015 to two groups.

The researchers included patients aged between 18 and 65 years old who underwent elective major abdominal surgery into random allocation. Patients were excluded if had a history of pulmonary disease and were unwilling or unable to take a deep breath effectively due to pain, diaphragmatic dysfunction, or opiate analgesia.

All study subjects were simple randomly allocated into the intervention and control groups according to the randomization table. The intervention group (23 subjects) received respiratory exercise with incentive spirometry before surgery, and the control group (23 subjects) were given standard preoperative care.

Subjects in the intervention group were trained to perform 15 minutes of respiratory exercise with incentive spirometry four times a day for two days before surgery by trained medical personnel. First, subjects were instructed to make a good seal over the incentive spirometry mouthpiece with their lips. Afterward, The subjects were asked to inhale deeply and slowly, and were also directed to hold their breath at the end of inspiration.

With alpha of 5%, beta of 10%, 39% postoperative pulmonary complication rate, as mentioned in the previous study,13 and assumption of that incentive spirometry can reduce the PPC to 30%, this study required at least 23 subjects in each group to see the effectiveness of using incentive spirometry before surgery in preventing PPC.

Measures In the intervention group, pulmonary function (vital capacity [VC], vital functional capacity [VFC], and Forced expiratory volume in the first second [FEV1]) were measured three times: two times before surgery (first day before undergoing the incentive spirometry procedure and second day after using the incentive spirometry) and one time after surgery. The control group measured pulmonary function three times: two times before surgery (on the first day of admission, on the day before surgery) and one time after surgery. In addition, postoperative pulmonary function was measured up to seven days following abdominal surgery, depending on the patient's ability.

On the first day after surgery, all subjects were examined by a pulmonologist, supplemented with a chest x-ray and blood gas analysis to assess the occurrence of postoperative pulmonary complications. PPC in this study included atelectasis (lung volume diminishing, caused by inadequate expansion of air cavity within lung parenchyma), pneumonia (all kinds of lung infection), and hypoxemia (ratio of PaO2: FiO2 less than 300).

The researchers used means (standard deviation, SD) and numbers (percentage,%) to describe the baseline subjects demographic and clinical characteristics. Henceforth, The researchers compared the change in lung function before and after surgery between intervention and control groups. An unpaired T-test was conducted to determine if the data were normally distributed. Alternatively, the Mann-Whitney test was done for abnormally distributed data. The researchers analyzed the comparison of lung complication incidence between experimental and control groups using chi-square or Fisher's exact test method. In this study, The researchers investigated the lung function of the experimental group before and after the incentive spirometry procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing major abdominal surgery
* aged between 18 and 65 years old
* Sign research informed consent

Exclusion Criteria:

* Emergency surgery
* Have a history of lung disorders
* Refusing to continue incentive spirometry
* Patients who cannot follow instructions in using the device incentive spirometry.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2015-08-10 (Actual); Study Completion 2015-09-01 (Actual)

PRIMARY OUTCOMES:
number of participants with atelectasis | day 1 until day 7
  The loss of lung volume is caused by inadequate expansion of the air spaces lung parenchyma. Assess based on plain chest X-rays examined by radiology and clinical assessment of a pulmonologist
number of participants with pneumonia | day 1 until day 7
  Any form of infection of the lung parenchyma. Assess based on plain chest X-rays examined by radiology and clinical assessment of a pulmonologist
number of participants with hypoxaemia | day 1 until day 7
  Hypoxaemia was defined as PaO2/FiO2 <300 as assessed by blood gas analysis

SECONDARY OUTCOMES:
vital capacity | Preoperative, day 1 before surgery, and until day 7 after surgery
  It is the total amount of air exhaled after maximal inhalation
forced vital capacity | Preoperative, day 1 before surgery, and until day 7 after surgery
  the maximum amount of air you can forcibly exhale from your lungs after fully inhaling
Forced expiratory volume in the first second | Preoperative, day 1 before surgery, and until day 7 after surgery
  the volume of air (in liters) exhaled in the first second during forced exhalation after maximal inspiration

IPD SHARING:
Plan to Share IPD: No
The data in this study cannot be shared because the research database is no longer available due to damage to the hard disk where the data is stored.

REFERENCES:
- [Background] McAlister FA, Bertsch K, Man J, Bradley J, Jacka M. Incidence of and risk factors for pulmonary complications after nonthoracic surgery. Am J Respir Crit Care Med. 2005 Mar 1;171(5):514-7. doi: 10.1164/rccm.200408-1069OC. Epub 2004 Nov 24. PMID 15563632
- [Background] Hall JC, Tarala RA, Hall JL, Mander J. A multivariate analysis of the risk of pulmonary complications after laparotomy. Chest. 1991 Apr;99(4):923-7. doi: 10.1378/chest.99.4.923. PMID 2009796
- [Background] Kodra N, Shpata V, Ohri I. Risk Factors for Postoperative Pulmonary Complications after Abdominal Surgery. Open Access Maced J Med Sci. 2016 Jun 15;4(2):259-63. doi: 10.3889/oamjms.2016.059. Epub 2016 May 22. PMID 27335597
- [Background] Kehrer HE. [Infantile autism and drug therapy]. Bibl Psychiatr. 1978;(157):91-7. No abstract available. German. PMID 348194
- [Background] Branson RD. The scientific basis for postoperative respiratory care. Respir Care. 2013 Nov;58(11):1974-84. doi: 10.4187/respcare.02832. PMID 24155356
- [Background] Haines KJ, Skinner EH, Berney S; Austin Health POST Study Investigators. Association of postoperative pulmonary complications with delayed mobilisation following major abdominal surgery: an observational cohort study. Physiotherapy. 2013 Jun;99(2):119-25. doi: 10.1016/j.physio.2012.05.013. Epub 2012 Sep 23. PMID 23219632
- [Background] Levy MM, Fink MP, Marshall JC, Abraham E, Angus D, Cook D, Cohen J, Opal SM, Vincent JL, Ramsay G; SCCM/ESICM/ACCP/ATS/SIS. 2001 SCCM/ESICM/ACCP/ATS/SIS International Sepsis Definitions Conference. Crit Care Med. 2003 Apr;31(4):1250-6. doi: 10.1097/01.CCM.0000050454.01978.3B. PMID 12682500
- [Background] Lyager S, Wernberg M, Rajani N, Boggild-Madsen B, Nielsen L, Nielsen HC, Andersen M, Moller J, Silberschmid M. Can postoperative pulmonary conditions be improved by treatment with the Bartlett-Edwards incentive spirometer after upper abdominal surgery? Acta Anaesthesiol Scand. 1979 Aug;23(4):312-9. doi: 10.1111/j.1399-6576.1979.tb01456.x. PMID 495034
- [Result] Patel K, Hadian F, Ali A, Broadley G, Evans K, Horder C, Johnstone M, Langlands F, Matthews J, Narayan P, Rallon P, Roberts C, Shah S, Vohra R. Postoperative pulmonary complications following major elective abdominal surgery: a cohort study. Perioper Med (Lond). 2016 May 23;5:10. doi: 10.1186/s13741-016-0037-0. eCollection 2016. PMID 27222707
- [Result] Yang CK, Teng A, Lee DY, Rose K. Pulmonary complications after major abdominal surgery: National Surgical Quality Improvement Program analysis. J Surg Res. 2015 Oct;198(2):441-9. doi: 10.1016/j.jss.2015.03.028. Epub 2015 Mar 18. PMID 25930169
- [Result] Kim TH, Lee JS, Lee SW, Oh YM. Pulmonary complications after abdominal surgery in patients with mild-to-moderate chronic obstructive pulmonary disease. Int J Chron Obstruct Pulmon Dis. 2016 Nov 9;11:2785-2796. doi: 10.2147/COPD.S119372. eCollection 2016. PMID 27877032
- [Result] Avila AC, Fenili R. Incidence and risk factors for postoperative pulmonary complications in patients undergoing thoracic and abdominal surgeries. Rev Col Bras Cir. 2017 May-Jun;44(3):284-292. doi: 10.1590/0100-69912017003011. English, Portuguese. PMID 28767805
- [Result] Carvalho CR, Paisani DM, Lunardi AC. Incentive spirometry in major surgeries: a systematic review. Rev Bras Fisioter. 2011 Sep-Oct;15(5):343-50. doi: 10.1590/s1413-35552011005000025. Epub 2011 Oct 14. PMID 22002191
- [Result] Thomas JA, McIntosh JM. Are incentive spirometry, intermittent positive pressure breathing, and deep breathing exercises effective in the prevention of postoperative pulmonary complications after upper abdominal surgery? A systematic overview and meta-analysis. Phys Ther. 1994 Jan;74(1):3-10; discussion 10-6. doi: 10.1093/ptj/74.1.3. PMID 8265725
- [Result] Tyson AF, Kendig CE, Mabedi C, Cairns BA, Charles AG. The effect of incentive spirometry on postoperative pulmonary function following laparotomy: a randomized clinical trial. JAMA Surg. 2015 Mar 1;150(3):229-36. doi: 10.1001/jamasurg.2014.1846. PMID 25607594
- [Result] Ramirez-Sarmiento A, Orozco-Levi M, Guell R, Barreiro E, Hernandez N, Mota S, Sangenis M, Broquetas JM, Casan P, Gea J. Inspiratory muscle training in patients with chronic obstructive pulmonary disease: structural adaptation and physiologic outcomes. Am J Respir Crit Care Med. 2002 Dec 1;166(11):1491-7. doi: 10.1164/rccm.200202-075OC. Epub 2002 Jul 19. PMID 12406842
- [Result] Kulkarni SR, Fletcher E, McConnell AK, Poskitt KR, Whyman MR. Pre-operative inspiratory muscle training preserves postoperative inspiratory muscle strength following major abdominal surgery - a randomised pilot study. Ann R Coll Surg Engl. 2010 Nov;92(8):700-7. doi: 10.1308/003588410X12771863936648. Epub 2010 Jul 26. PMID 20663275
- [Result] Toor H, Kashyap S, Yau A, Simoni M, Farr S, Savla P, Kounang R, Miulli DE. Efficacy of Incentive Spirometer in Increasing Maximum Inspiratory Volume in an Out-Patient Setting. Cureus. 2021 Oct 4;13(10):e18483. doi: 10.7759/cureus.18483. eCollection 2021 Oct. PMID 34754645
- [Result] Kotani T, Akazawa T, Sakuma T, Nagaya S, Sonoda M, Tanaka Y, Katogi T, Nemoto T, Minami S. Effects of Incentive Spirometry on Respiratory Motion in Healthy Subjects Using Cine Breathing Magnetic Resonance Imaging. Ann Rehabil Med. 2015 Jun;39(3):360-5. doi: 10.5535/arm.2015.39.3.360. Epub 2015 Jun 30. PMID 26161341
- [Result] Kulnik ST, Rafferty GF, Birring SS, Moxham J, Kalra L. A pilot study of respiratory muscle training to improve cough effectiveness and reduce the incidence of pneumonia in acute stroke: study protocol for a randomized controlled trial. Trials. 2014 Apr 12;15:123. doi: 10.1186/1745-6215-15-123. PMID 24725276
- [Result] do Nascimento Junior P, Modolo NS, Andrade S, Guimaraes MM, Braz LG, El Dib R. Incentive spirometry for prevention of postoperative pulmonary complications in upper abdominal surgery. Cochrane Database Syst Rev. 2014 Feb 8;2014(2):CD006058. doi: 10.1002/14651858.CD006058.pub3. PMID 24510642